CLINICAL TRIAL: NCT01753739
Title: A Dose-Ranging Study to Evaluate the Safety and Efficacy of Bepotastine Besilate Nasal Sprays in the Treatment of Seasonal Allergic Rhinitis (SAR) in Subjects With a Demonstrated History of Mountain Cedar Pollen Allergic Sensitivity
Brief Title: Bepotastine Besilate Nasal Sprays in the Treatment of Seasonal Allergic Rhinitis (SAR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 823
Record Dates: First submitted 2012-12-18; First posted 2012-12-20 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — bepotastine besilate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Bepotastine besilate Concentration 1 (Experimental): Bepotastine besilate nasal spray, BID for 14 days.
  Interventions: Drug: Bepotastine besilate
- Placebo (Active Comparator): Placebo nasal spray BID for 14 days
  Interventions: Drug: Placebo
- Bepotastine besilate Concentration 2 (Experimental): Bepotastine besilate nasal spray, BID for 14 days.
  Interventions: Drug: Bepotastine besilate
- Bepotastine besilate Concentration 3 (Experimental): Bepotastine besilate nasal spray, BID for 14 days.
  Interventions: Drug: Bepotastine besilate
- Bepotastine besilate Concentration 4 (Experimental): Bepotastine besilate nasal spray, BID for 14 days.
  Interventions: Drug: Bepotastine besilate

INTERVENTIONS:
Drug: Bepotastine besilate — Nasal spray administered in the morning and at night approximately 12 hours apart daily for 14 days
  Arms: Bepotastine besilate Concentration 1; Bepotastine besilate Concentration 2; Bepotastine besilate Concentration 3; Bepotastine besilate Concentration 4
Drug: Placebo — Nasal spray administered in the morning and at night approximately 12 hours apart daily for 14 days
  Arms: Placebo

SUMMARY:
This study will examine dose ranging characteristics of bepotastine besilate nasal spray compared to placebo nasal spray in 600 male or female subjects 12 years of age and older with active seasonal allergic rhinitis (SAR) and a demonstrated history of allergic sensitivity to Mountain Cedar pollen for at least 2 years prior to the study.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a male or female 12 years of age or older.
* Have a documented history of SAR resulting from exposure to Mountain Cedar pollen for a minimum of 2 years immediately preceding Screening Visit 1.
* Have demonstrated sensitivity to Mountain Cedar pollen through a standard skin prick test.
* Have a minimum rTNSS of at least 6 units for the morning (AM) assessment on the day of Visit 2 and Visit 3.
* Have a minimum average rTNSS score of at least 6 units for 3 of the worst 4 days prior to Visit 3 plus the AM assessment on the day of Visit 3.
* Have a minimum stuffy nose score of at least 2 units on the day of Visit 3.
* Have a minimum average stuffy nose score of at least 2 units for 3 of the worst 4 days prior to Visit 3 plus the AM assessment on the day of Visit 3.
* Have at least one score ≥ 2 units at Visit 3 of any of the RQLQ(S) questions #4-#6 regarding sleep.

Exclusion Criteria:

* Have a nasal condition which, in the opinion of the Investigator, interferes with successful nasal drug administration or absorption (in either nostril) within the last 60 days prior to Screening Visit 2.
* Have asthma requiring medication other than intermittent use of an inhaled short-acting β-agonist.
* Is participating or have participated in any investigational drug or device study within 30 days preceding Visit 2.
* Have had nasal or sinus surgery within 12 weeks of Visit 2.
* Have a known sensitivity to bepotastine besilate or any excipient component of the investigational product (IP).
* For female subjects 12 years of age or older (other than those who have been menopausal for at least 24 months or those who are surgically sterile), are pregnant, planning to become pregnant, or nursing/lactating, or refuses to abide by the contraception stipulations in the inclusion criteria.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Williams, Ph.D., Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bepotastine Besilate 0.5%; Bepotastine Besilate 1%; Bepotastine Besilate 2%; Bepotastine Besilate 4%: Bepotastine besilate nasal spray, BID for 14 days.
  Bepotastine besilate: Nasal spray administered in the morning and at night approximately 12 hours apart daily for 14 days
Period: Overall Study
Arm/Group | Placebo | Bepotastine Besilate 0.5% | Bepotastine Besilate 1% | Bepotastine Besilate 2% | Bepotastine Besilate 4%
Started | 124 | 123 | 123 | 124 | 123
Completed | 120 | 118 | 118 | 117 | 120
Not Completed | 4 | 5 | 5 | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bepotastine Besilate 0.5% | Bepotastine Besilate 1% | Bepotastine Besilate 2% | Bepotastine Besilate 4% | Total
Number analyzed (Participants) | 124 | 123 | 123 | 124 | 123 | 617
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (14.7) | 41.3 (15.5) | 41.3 (14.7) | 42.4 (15.1) | 39.8 (14.6) | 41.3 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 74 | 81 | 77 | 73 | 381
  Male | 48 | 49 | 42 | 47 | 50 | 236

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline (Pre-Dose) Twice Daily Averaged Subject-rated Reflective Total Nasal Symptom Score (TNSS)
Description: Total nasal symptom score (TNSS) was the summed scores for nasal pruritus [itching], rhinorrhea [runny nose], nasal congestion, and sneezing. Individual nasal symptoms were each rated on a 4-point scale from 0-3 (0=Absent, 1=Mild, 2=Moderate, 3=Severe), with no half-unit assessments. TNSS was the sum score of 4 nasal symptoms with a minimum score of 0 units and a maximum score of 12 units, with higher score corresponding to increased nasal allergy symptoms. Morning and evening scores were averaged.
Time Frame: 14 Days
Population: The analysis population included randomized participants who had received at least 1 dose of study drug. There was no imputation of missing data at Day 14.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Bepotastine Besilate 0.5% | Bepotastine Besilate 1% | Bepotastine Besilate 2% | Bepotastine Besilate 4%
Number analyzed (Participants) | 122 | 121 | 122 | 122 | 123
score on a scale | -1.19 (2.22) | -1.58 (2.28) | -1.68 (2.24) | -1.63 (2.21) | -1.55 (2.23)

2. Secondary Outcome: Mean Change From Baseline (Pre-Dose) in Morning Averaged Subject-rated Reflective (TNSS)
Description: Total nasal symptom score (TNSS) was the summed scores for nasal pruritus [itching], rhinorrhea [runny nose], nasal congestion, and sneezing. Individual nasal symptoms were each rated on a 4-point scale from 0-3 (0=Absent, 1=Mild, 2=Moderate, 3=Severe), with no half-unit assessments. TNSS was the sum score of 4 nasal symptoms with a minimum score of 0 units and a maximum score of 12 units, with higher score corresponding to increased nasal allergy symptoms.
Time Frame: 14 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Bepotastine Besilate 0.5% | Bepotastine Besilate 1% | Bepotastine Besilate 2% | Bepotastine Besilate 4%
Number analyzed (Participants) | 122 | 121 | 122 | 122 | 123
score on a scale | -1.29 (2.28) | -1.68 (2.35) | -1.72 (2.22) | -1.71 (2.31) | -1.66 (2.31)

3. Secondary Outcome: Mean Change From Baseline (Pre-Dose) in Evening Averaged Subject-rated Reflective Total Nasal Symptom Score (TNSS)
Description: as for outcome 2
Time Frame: 14 Days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Bepotastine Besilate 0.5% | Bepotastine Besilate 1% | Bepotastine Besilate 2% | Bepotastine Besilate 4%
Number analyzed (Participants) | 122 | 121 | 122 | 122 | 123
score on a scale | -1.14 (2.24) | -1.55 (2.34) | -1.70 (2.33) | -1.60 (2.23) | -1.50 (2.25)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Placebo | Bepotastine Besilate 0.5% | Bepotastine Besilate 1% | Bepotastine Besilate 2% | Bepotastine Besilate 4%
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/123 | 0/123 | 0/124 | 0/123
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/123 | 0/123 | 0/124 | 0/123
Other Adverse Events (participants affected / at risk) | 1/124 | 8/123 | 12/123 | 15/124 | 18/123
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=124) | Bepotastine Besilate 0.5% (N=123) | Bepotastine Besilate 1% (N=123) | Bepotastine Besilate 2% (N=124) | Bepotastine Besilate 4% (N=123)
Mild taste following instillation (General disorders) | 1 | 8 | 12 | 15 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.